CLINICAL TRIAL: NCT05126043
Title: Triglyceride/High Density Lipoprotein-cholesterol Ratio as a Novel Marker of Atherosclerosis in Patients With Acute Coronary Syndrome
Brief Title: Lipid Profile in Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fatma mohamed Ahmed Anwer, Principal investigator, Sohag University
Other Study IDs: Acute coronary syndrome
Record Dates: First submitted 2021-11-05; First posted 2021-11-18 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Triglycerides/high density lipoprotein ratio — Lipid profile

SUMMARY:
This study aims to assess the TG/Hdl-c ratio in patients with acute coronary syndrome as a novel marker of atherosclerosis.

DETAILED DESCRIPTION:
Cross sectional study to:

assess triglycerides/high density lipoprotein-cholesterol ratio as a novel atherogenic marker in patients presenting with acute coronary syndrome

ELIGIBILITY:
Inclusion Criteria:

* all patients presented with acute coronary syndrome

Exclusion Criteria:

* patients less than 18 years
* rheumatic heart disease
* congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presented with acute coronary syndrome admitted to coronary care unit of Sohag University hospital according to inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Coronary care unit admission | From date of randomization up to 1 month
  Acute coronary syndrome hospitalization and cardiovascular deathes and estimated hazar ratios (HR) by use of multivariable Cox regression models

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Ahmed, Lecturer, Study Chair — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Dzubur A, Ejubovic M, Fajkic A, Dervisevic A, Durak Nalbantic A, Avdic Agic A, Dzubur A, Mekic M. The serum triglyceride to high-density lipoprotein (HDL) ratio in patients with acute coronary syndrome with and without renal dysfunction. Med Glas (Zenica). 2019 Feb 1;16(1):28-34. doi: 10.17392/990-19. PMID 30680982